# **INFORMED CONSENT FORM** (for Participation in a Clinical Trial)

Official Study Title:

Is The Level of Muscle Damage After The Drop Jump Protocol Affected By Body Weight and BMI?

NCT Number:

(Not yet assigned – to be updated upon registration)

Document Date: October 15, 2024

Principal Investigator:
Dr. Melike Nur EROGLU
Sakarya University of Applied Sciences
Email: melikeeroglu@subu.edu.tr

Phone: +90 5384982024

**Study Location:** 

Tokat Gaziosmanpaşa University, Faculty of Sports Sciences

This document provides information about the clinical study mentioned above. Your participation is entirely voluntary. Please read this form carefully before deciding to take part.

# 1. Introduction and Purpose of the Study

You are being invited to participate in a scientific research study. The purpose of this study is to investigate whether muscle damage induced by a drop jump (DJ) protocol varies based on participants' body weight and body mass index (BMI).

#### 2. Procedures

If you agree to participate:

- You will perform a drop jump exercise consisting of 100 jumps from a 60 cm platform, performed in 5 sets.
- You will provide blood samples at three time points: before the exercise, immediately after, and 24 hours later.
- The blood samples will be analyzed for biomarkers such as Creatine Kinase (CK) and Lactate Dehydrogenase (LDH).
- The total duration of participation is approximately 2 days.

#### 3. Potential Risks and Discomforts

- Muscle soreness, stiffness, or fatigue may occur after the drop jump protocol.
- Bruising or mild discomfort may occur at the blood draw site.

#### 4. Potential Benefits

There is no direct personal benefit; however, your participation will contribute to the understanding of how body weight influences exercise-induced muscle damage.

## 5. Confidentiality

All personal and health information will remain confidential. Your identity will not be revealed in any publication resulting from this study. Data will be stored securely and only accessible to authorized research personnel.

## 6. Voluntary Participation

Your participation is completely voluntary. You may withdraw at any time without any penalty or loss of benefits.

# 7. Questions

If you have any questions about the study or your rights as a participant, you may contact the principal investigator or the ethics committee of Tokat Gaziosmanpaşa University.

# 8. Consent

Participant Statement:

I have read and understood the information above. I have had the opportunity to ask questions and have received satisfactory answers. I voluntarily agree to participate in this study.

| Name of Participant: |
|-------------------------------|
| Signature of Participant: |
| Date: |
| Name of Researcher (Witness): |
| Signature of Researcher: |
| Dota |